CLINICAL TRIAL: NCT05474391
Title: The Value of MammaPrint in Adjuvant Therapy Decision Among Pre-menopausal Breast Cancer Patients: a Survey Based on Clinical Staff
Brief Title: MammaPrint Value for Pre-menopausal Breast Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-16
Record Dates: First submitted 2022-07-22; First posted 2022-07-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MammaPrint group: Pre-menopausal breast cancer patients received MammaPrint test.

SUMMARY:
Nearly 200 cases are to be enrolled. The information of patient age, histologic grade, tumor size, ER and PR status, Ki-67 index, surgery mode should be provided. The adjuvant therapy regime (chemotherapy: none, TC*4, TC*6 or EC-T; endocrine therapy: TAM, OFS+TAM, OFS+AI) will be compared before and after MammaPrint testing. About 20 clinical staffs are enrolled to participate in this survey for the clinical decision making. Each case could be chosen five times at random.

ELIGIBILITY:
Inclusion Criteria:

1. pre-menopausal breast cancer patients aged less than 50 years old.
2. Pathology confirmed invasive dutal carcinoma or invasive lobular carcinoma.
3. receiving breast conserving surgery or mastectomy with/without reconstruction; sentinel lymph node biopsy or axillary lymph node dissection.
4. TNM staging: T1b-T2N0-1M0.
5. molecular subtype: ER positive/HER2 negative.
6. MammaPrint testing before initiation of adjuvant therapy.

Exclusion Criteria:

1. Incomplete medical history.
2. Pregnancy or lactation.
3. Contradiction of chemotherapy or ovarian function suppression.

Max Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with breast cancer (according to ICD-10)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Treatment decision survey | 6 weeks
  Treatment decision change after MammaPrint testing

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided